CLINICAL TRIAL: NCT00834782
Title: Comparison of Pascal Dynamic Contour Tonometer, Reichart Ocular Response Analyzer and Goldmann Applanation Tonometer in Eyes After Penetrating Keratoplasty
Brief Title: Comparison of DCT, ORA and GAT in Eyes After Penetrating Keratoplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr Ido Didi Fabian, Sheba Medical Center, Goldschleger eye institute
Other Study IDs: SHEBA-09-6902-IDF-CTIL
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Corneal Transplantation
Keywords: PK; IOP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IOP: Measuring IOP
  Interventions: Procedure: IOP measurement

INTERVENTIONS:
Procedure: IOP measurement — Measuring IOP

SUMMARY:
To compare intraocular pressure (IOP) measured by the Reichert Ocular Response Analyzer (ORA), Pascal dynamic contour tonometer (DCT) and Goldmann applanation tonometer (GAT) in eyes after Penetrating Keratoplasty (KPL)

DETAILED DESCRIPTION:
A few tonometers are used today in clinical practice for measuring intra ocular pressure (IOP). Each tonometer is based on different technology.

Post penetrating keratoplasty (PK) eyes are at risk for developing secondary glaucoma (9-14%). Elevation of the IOP may cause rejection of the graft or alternately a loss in the endothelial cell layer count causing decompensation of the cornea. Therefore, measuring accurately the IOP in this population is of great importance.

Measuring IOP in post PK is not an easy challenge, mainly because of parameters like the central corneal thickness (CCT), the curvature of the cornea, the axial length and biomechanical properties which diverse from normal eyes.

The Goldmann applanation tonometer (GAT) is the gold standard tonometer for measuring IOP and is the most popular tonometer clinically used. IOP measurements via the GAT are based on the assumption that the CCT is constant. post PK eyes CCT might diverse from normal eyes causing GAT IOP measurements to be inaccurate. The Pascal dynamic contour tonometer (DCT) measures IOP independently of corneal parameters. The Ocular response analyzer (ORA) is based on a non contact technique of measurement. The tonometer is thought to be independent of factors such as CCT.

The aim of the study is to compare intraocular pressure (IOP) measured by the Reichert Ocular Response Analyzer (ORA), Pascal dynamic contour tonometer (DCT) and Goldmann applanation tonometer (GAT) in eyes after Penetrating Keratoplasty (KPL). In addition its aim is to discover the dependence of different parameters, like - CCT, curvature of the cornea, axial length and biomechanical properties on IOP measurement to elucidate the appropriate tonometer for this population.

ELIGIBILITY:
Inclusion Criteria:

* Eyes after KPL surgery at the Goldschleger Eye Institute in the last 10 years.

Exclusion Criteria:

* Uncooperative subjects for whom good quality results are unattainable.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients post keratoplasty surgery
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-12 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Intra ocular pressure | 1 year

SECONDARY OUTCOMES:
Corneal compensated intra ocular pressure, Corneal hysteresis, Corneal resistance factor | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Melamed, Prof, Study Chair — Sheba medical center, head of Sam rotberg glaucoma center
Locations (2):
- Israel (2):
  - Goldschleger eye institute, Sheba medical center, Ramat Gan
  - The Goldschleger eye institute, Sheba Medical Center, Tel Aviv University, Ramat Gan

REFERENCES:
- [Background] Congdon NG, Broman AT, Bandeen-Roche K, Grover D, Quigley HA. Central corneal thickness and corneal hysteresis associated with glaucoma damage. Am J Ophthalmol. 2006 May;141(5):868-75. doi: 10.1016/j.ajo.2005.12.007. Epub 2006 Mar 9. PMID 16527231
- [Background] Jain AK, Saini JS, Gupta R. Tonometry in normal and scarred corneas, and in postkeratoplasty eyes: a comparative study of the Goldmann, the ProTon and the Schiotz tonometers. Indian J Ophthalmol. 2000 Mar;48(1):25-32. PMID 11271930
- [Background] Kerautret J, Colin J, Touboul D, Roberts C. Biomechanical characteristics of the ectatic cornea. J Cataract Refract Surg. 2008 Mar;34(3):510-3. doi: 10.1016/j.jcrs.2007.11.018. PMID 18299080
- [Background] Luce DA. Determining in vivo biomechanical properties of the cornea with an ocular response analyzer. J Cataract Refract Surg. 2005 Jan;31(1):156-62. doi: 10.1016/j.jcrs.2004.10.044. PMID 15721708
- [Background] Medeiros FA, Weinreb RN. Evaluation of the influence of corneal biomechanical properties on intraocular pressure measurements using the ocular response analyzer. J Glaucoma. 2006 Oct;15(5):364-70. doi: 10.1097/01.ijg.0000212268.42606.97. PMID 16988597
- [Background] Mollan SP, Wolffsohn JS, Nessim M, Laiquzzaman M, Sivakumar S, Hartley S, Shah S. Accuracy of Goldmann, ocular response analyser, Pascal and TonoPen XL tonometry in keratoconic and normal eyes. Br J Ophthalmol. 2008 Dec;92(12):1661-5. doi: 10.1136/bjo.2007.136473. Epub 2008 Aug 29. PMID 18757471
- [Background] Pandav SS, Sharma A, Gupta A, Sharma SK, Gupta A, Patnaik B. Reliability of proton and goldmann applanation tonometers in normal and postkeratoplasty eyes. Ophthalmology. 2002 May;109(5):979-84. doi: 10.1016/s0161-6420(02)00974-0. PMID 11986107
- [Background] Rao VJ, Gnanaraj L, Mitchell KW, Figueiredo FC. Clinical comparison of ocular blood flow tonometer, Tonopen, and Goldmann applanation tonometer for measuring intraocular pressure in postkeratoplasty eyes. Cornea. 2001 Nov;20(8):834-8. doi: 10.1097/00003226-200111000-00011. PMID 11685061
- [Background] Touboul D, Roberts C, Kerautret J, Garra C, Maurice-Tison S, Saubusse E, Colin J. Correlations between corneal hysteresis, intraocular pressure, and corneal central pachymetry. J Cataract Refract Surg. 2008 Apr;34(4):616-22. doi: 10.1016/j.jcrs.2007.11.051. PMID 18361984